CLINICAL TRIAL: NCT03824769
Title: Is Long-term Maintenance Worth the Wait? Using Real Time Data Capture to Examine Delayed Discounting as a Putative Target of Physical Activity Adherence in Weight Loss Maintenance Interventions
Brief Title: Physical Activity Choices Everyday
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University at Buffalo (Other); Kent State University (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Amy Gorin, Director, Institute for Collaboration on Health, Intervention, and Policy Professor, Psychological Sciences, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-153; R21NR018359 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: Weight Loss Maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss Maintenance + Healthy Thinking (Active Comparator): Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
  Interventions: Behavioral: Weight Loss Maintenance + Healthy Thinking
- Behavioral Weight Loss Maintenance Treatment + Future Thinking (Experimental): Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
  Interventions: Behavioral: Weight Loss Maintenance Treatment + Future Thinking

INTERVENTIONS:
Behavioral: Weight Loss Maintenance + Healthy Thinking — Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
  Arms: Behavioral Weight Loss Maintenance + Healthy Thinking
Behavioral: Weight Loss Maintenance Treatment + Future Thinking — Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
  Arms: Behavioral Weight Loss Maintenance Treatment + Future Thinking

SUMMARY:
This study aims to test two strategies for weight loss maintenance. It involves two phases, a weight loss phase and a maintenance phase. During Phase I (the weight loss phase), participants will receive a 16-week, Web-based behavioral weight loss program that involves access to weekly weight loss information and weekly personalized feedback on diet, activity, and weight loss goals. Individuals who lose at least 5% of their initial body weight during this program, will be invited to participate in Phase II. During Phase II, two 4-month treatments for weight loss maintenance will be tested. At the beginning of Phase II, participants will be randomly assigned to one of the two maintenance programs: (1) a behavioral maintenance program that involves in-person group meetings plus daily exercises in which information about a healthy lifestyle is reviewed or (2) a behavioral maintenance program that involves in-person group meetings plus daily exercises in which descriptions of positive future events are reviewed. Throughout the study, participants will complete assessments that examine the effects of the interventions on delay discounting, physical activity, weight, and other important health and psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70
* Body Mass Index between 30-50
* English Speaking
* Have a smartphone that can be used for study activities

Exclusion Criteria:

* Report being unable to walk 2 blocks without stopping
* Are currently participating in weight loss treatment, have a history of bariatric surgery, or lost ≥5% in the past 6-months
* Are pregnant or plan to become pregnant within 1 year
* Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that could jeopardize their safety in a weight control program with diet and exercise guidelines
* History of or current traumatic brain injury, dementia or Alzheimer's disease; a history of Multiple Sclerosis, or other neurological disorders
* Report conditions that, in the judgment of the PI, would render them unlikely to follow the protocol (e.g., relocation, dementia, unable to read and write in English)
* Have no Internet access or unwilling to use personal smartphone for study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gorin, PhD, Principal Investigator — University of Connecticut
Locations (1):
- UConn Weight Management Research Laboratory, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leahey TM, Gorin AA, Wyckoff E, Denmat Z, O'Connor K, Field C, Dunton GF, Gunstad J, Huedo-Medina TB, Gilder C. Episodic future thinking, delay discounting, and exercise during weight loss maintenance: The PACE trial. Health Psychol. 2020 Sep;39(9):796-805. doi: 10.1037/hea0000860. PMID 32833481

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, participants began Phase I, a 16-week weight loss program aiming to induce clinically significant weight loss (5% of starting body weight). After Phase I, eligibility to continue to Phase II (weight maintenance) was evaluated. Those who lost at least 5% of their body weight remained eligible. Given that Phase II was the primary focus of the study, primary outcome data were analyzed only from randomized, Phase II participants (eligible subset of Phase I participants).
Groups:
- Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
  All participants randomized to this treatment arm completed Phase I (Weight Loss Phase) and were eligible for Phase II (Weight Maintenance Phase).
- Phase II (RCT): Behavioral Weight Loss Maintenance Treatment + Future Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
  Weight Loss Maintenance Treatment + Future Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
- Phase I Only (Weight Loss Phase): 16 Weeks: This group consists of the participants who enrolled in Phase I (Weight Loss Phase) but were not randomized to Phase I because they dropped out or were not eligible for Phase II (Weight Maintenance Phase).
Period: Phase I (Weight Loss): 16 Weeks
Arm/Group | Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking | Phase II (RCT): Behavioral Weight Loss Maintenance Treatment + Future Thinking | Phase I Only (Weight Loss Phase): 16 Weeks
Started | 24 | 28 | 108
Completed | 24 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. All participants in this arm were eligible and randomized into the Phase II Weight Maintenance RCT.) | 28 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. All participants in this arm were eligible and randomized into the Phase II Weight Maintenance RCT.) | 0 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. Because participants in this group did not meet all 3 of these requirements and were not randomized, all are considered incomplete.)
Not Completed | 0 | 0 | 108
Period: Phase II (Weight Maintenance): 4 Months
Arm/Group | Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking | Phase II (RCT): Behavioral Weight Loss Maintenance Treatment + Future Thinking | Phase I Only (Weight Loss Phase): 16 Weeks
Started | 24 | 28 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
1 Month Assessment | 22 | 27 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
2 Month Assessment | 21 | 26 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
Completed | 22 | 28 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Weight Loss Maintenance + Healthy Thinking | Behavioral Weight Loss Maintenance Treatment + Future Thinking | Phase I Only (Weight Loss Phase): 16 Weeks | Total
Number analyzed (Participants) | 24 | 28 | 108 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.83 (10.26) | 48.11 (13.02) | 46.80 (12.03) | 46.88 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 96 | 138
  Male | 3 | 7 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 14 | 17
  Not Hispanic or Latino | 21 | 28 | 94 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Black or African American | 3 | 0 | 24 | 27
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  White | 19 | 24 | 73 | 116
  More than One Race | 2 | 0 | 4 | 6
  Other | 0 | 1 | 1 | 2
  Prefer not to answer | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 108 | 160
Weekly Moderate-Vigorous Physical Activity Minutes, Accelerometry [Mean (Standard Deviation); unit: minutes] — Weekly minutes of moderate to vigorous physical activity measured via a waist worn accelerometer during the Phase II baseline assessment. At Phase II baseline, participants were instructed to wear the accelerometer on their right waist during all waking hours for 7 days. Participants with a minimum of 600 min per day of valid daily wear time for at least 4 days were included in reported outcomes. Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  minutes
    number analyzed (Participants) | 24 | 28 | 0 | 52
    (all) | 194.29 (119.595) | 229.82 (162.393) |  | 213.42 (143.985)
Delay Discounting (Adjusting Amount Task) [Mean (Standard Deviation); unit: k-value] — Baseline delay discounting measured using the Adjusting Amount task during the Phase II baseline assessment. Delay discounting refers to the decline in the present value of a reward with delay to its receipt. The Adjusting Amount task identifies an individual's discount rate, which reflects how much they devalue future rewards. Discount rate is represented by "k". A higher "k" value means a greater preference for immediate rewards and a higher devaluation of future rewards. Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  k-value
    number analyzed (Participants) | 24 | 28 | 0 | 52
    (all) | 0.002589348 (0.003302) | 0.021894643 (0.108428) |  | 0.012984507 (0.079520)
Delay Discounting (Monetary Choice Questionnaire) [Mean (Standard Deviation); unit: k-value] — Baseline delay discounting measured using the Monetary Choice Questionnaire (MCQ) task during the Phase II baseline assessment. Delay discounting refers to the decline in the present value of a reward with delay to its receipt. The MCQ task identifies an individual's discount rate, which reflects how much they devalue future rewards. Discount rate is represented by "k". A higher "k" value means a greater preference for immediate rewards and a higher devaluation of future rewards. Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  k-value
    number analyzed (Participants) | 24 | 28 | 0 | 52
    (all) | 0.017834 (0.019678) | 0.025506 (0.047832) |  | 0.021965 (0.037427)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  kilograms
    number analyzed (Participants) | 24 | 28 | 0 | 52
    (all) | 94.89 (17.09) | 92.00 (16.38) |  | 93.33 (16.61)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Moderate-Vigorous Physical Activity Minutes, Accelerometry
Description: Change in weekly minutes of moderate to vigorous physical activity measured via a waist worn accelerometer during the Phase II maintenance program. At each assessment time point, participants were instructed to wear the accelerometer on their right waist during all waking hours for 7 days. Participants with a minimum of 600 min of valid daily wear time for at least 4 days were included in reported outcomes.
Time Frame: Phase II baseline to 1 month, 2 months and 4 months (end of treatment)
Population: The number of participants analyzed in this outcome measure generally reflects the number that completed accelerometry assessment procedures at each timepoint. At the 2 month assessment, one Healthy Thinking participant's data was excluded due to insufficient device wear time. All other missing participant data indicates that the participant did not complete this assessment procedure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Behavioral Weight Loss Maintenance + Healthy Thinking | Behavioral Weight Loss Maintenance Treatment + Future Thinking
Number analyzed (Participants) | 24 | 28
Minutes
  Phase II baseline to 1-month: number analyzed (Participants) | 21 | 25
  Phase II baseline to 1-month | -21.4286 (61.52851) | -53.9600 (149.60712)
  Phase II baseline to 2-month: number analyzed (Participants) | 21 | 25
  Phase II baseline to 2-month | 19.6000 (100.36900) | -38.6800 (108.40846)
  Phase II baseline to 4-month: number analyzed (Participants) | 21 | 26
  Phase II baseline to 4-month | -12.7143 (96.02403) | -65.7308 (126.15627)

2. Primary Outcome: Delay Discounting (Adjusting Amount Task)
Description: Change in delay discounting measured using the Adjusting Amount task during the Phase II maintenance program. Delay discounting refers to the decline in the present value of a reward with delay to its receipt. The Adjusting Amount task identifies an individual's discount rate, which reflects how much they devalue future rewards. In the task, participants are presented with a choice between a smaller, immediate (hypothetical) monetary reward and a larger, delayed (hypothetical) monetary reward. Then, using a titration procedure, the delayed reward amount is adjusted based on the participant's choices to find the point at which they are indifferent between the two options (i.e., discounting rate). The discount rate is represented by "k". A higher "k" value means a steeper discount rate, indicating a greater preference for immediate rewards and a higher devaluation of future rewards.
Time Frame: Phase II baseline to 1 month, 2 months and 4 months (end of treatment)
Population: The number of participants analyzed in each group reflects the number of randomized participants that completed the delay discounting measure at each timepoint.
Measure: Mean (Standard Deviation); unit: k-value
Arm/Group | Behavioral Weight Loss Maintenance + Healthy Thinking | Behavioral Weight Loss Maintenance Treatment + Future Thinking
Number analyzed (Participants) | 24 | 28
k-value
  Baseline to 1-month: number analyzed (Participants) | 22 | 28
  Baseline to 1-month | 0.001280 (0.003962) | 0.107264 (0.547971)
  Baseline to 2-month: number analyzed (Participants) | 21 | 26
  Baseline to 2-month | 0.000165 (0.003824) | 0.108922 (0.558786)
  Baseline to 4-month: number analyzed (Participants) | 22 | 28
  Baseline to 4-month | -0.000071 (0.003989) | 0.101414 (0.538400)

3. Primary Outcome: Delay Discounting (Monetary Choice Questionnaire)
Description: Change in delay discounting measured using the Monetary Choice Questionnaire (MCQ) task during the Phase II maintenance program. Delay discounting refers to the decline in the present value of a reward with delay to its receipt. The MCQ identifies an individual's discount rate, which reflects how much they devalue future rewards. In the task, each question asks participants to make a choice between a smaller, immediate (hypothetical) monetary reward and a larger, delayed (hypothetical) reward. Unlike the Adjusting Amount task, each MCQ question includes different combinations of delay periods and reward amounts that are not influenced by previous responses (i.e., delay periods and reward amounts are static and the same for each participant). The discount rate is represented by "k". A higher "k" value means a steeper discount rate, indicating a greater preference for immediate rewards and a higher devaluation of future rewards.
Time Frame: Phase II baseline to 2 months and 4 months (end of treatment)
Population: The number of participants analyzed at each timepoint reflects the number of randomized participants who completed this measure.
Measure: Mean (Standard Deviation); unit: k-value
Arm/Group | Behavioral Weight Loss Maintenance + Healthy Thinking | Behavioral Weight Loss Maintenance Treatment + Future Thinking
Number analyzed (Participants) | 24 | 28
k-value
  Baseline to 2-months: number analyzed (Participants) | 21 | 26
  Baseline to 2-months | 0.002863 (0.029509) | -0.007161 (0.017930)
  Baseline to 4-months: number analyzed (Participants) | 22 | 26
  Baseline to 4-months | -0.001625 (0.022689) | -0.004049 (0.015750)

4. Secondary Outcome: Weight
Description: Weight change from end of Phase 1 weight loss program to end of Phase II maintenance program
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Behavioral Weight Loss Maintenance + Healthy Thinking | Behavioral Weight Loss Maintenance Treatment + Future Thinking
Number analyzed (Participants) | 22 | 28
kilograms | -11.87 (7.66) | -9.28 (6.63)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for all participants enrolled in Phase I (including participants randomized to Phase II) from from the start of the program to the post-Phase I assessment (a total of 16 weeks). For participants randomized to Phase II, Adverse events data were additionally collected at the Phase II baseline, 2-month and 4-month assessment visits (a total of 32 weeks).
Groups:
- Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
  Weight Loss Maintenance + Healthy Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will be asked to read short passages related to nutrition and a healthy lifestyle through our study website twice a day for the duration of treatment.
- Phase II (RCT) Behavioral Weight Loss Maintenance Treatment + Future Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
  Weight Loss Maintenance Treatment + Future Thinking: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive a 4-month behavioral weight maintenance intervention consisting of 7 sessions that focus on evidence-based weight management strategies focused on diet, exercise, and behavioral skills. In this treatment, participants will create descriptions of upcoming positive events and will be asked to read short passages through our study website at least twice a day for the duration of treatment.
Arm/Group | Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking | Phase II (RCT) Behavioral Weight Loss Maintenance Treatment + Future Thinking | Phase I Only (Weight Loss Phase): 16 Weeks
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28 | 2/108
Other Adverse Events (participants affected / at risk) | 9/24 | 7/28 | 4/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking (N=24) | Phase II (RCT) Behavioral Weight Loss Maintenance Treatment + Future Thinking (N=28) | Phase I Only (Weight Loss Phase): 16 Weeks (N=108)
Other (General disorders) | 0 | 0 | 1
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II (RCT): Behavioral Weight Loss Maintenance + Healthy Thinking (N=24) | Phase II (RCT) Behavioral Weight Loss Maintenance Treatment + Future Thinking (N=28) | Phase I Only (Weight Loss Phase): 16 Weeks (N=108)
Muscle or bone injury (e.g., broken bone, torn ligament, sprain) (Injury, poisoning and procedural complications) | 3 | 3 | 1
Other (General disorders) | 4 | 3 | 3
Gall bladder attack or surgery (Gastrointestinal disorders) | 1 | 0 | 0
New diagnosis, started treatment, or hospitalized for depression (Psychiatric disorders) | 0 | 1 | 0
Stroke, ministroke (TIA), or other neurological problems (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03824769/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03824769/ICF_001.pdf